CLINICAL TRIAL: NCT03869970
Title: Active Injury Management (AIM) After Pediatric Concussion
Acronym: AIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Danny Thomas, Associate Professor Pediatric Emergency Medicine, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO00033221
Record Dates: First submitted 2019-02-26; First posted 2019-03-11 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Brain Concussion
Keywords: Concussion
MeSH Terms: conditions — Brain Concussion | interventions — Exercise; Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Rest (Active Comparator): Discharge instructions focused on 24 - 48 hours of rest then symptom guided activity, Fitbit monitored.
  Interventions: Behavioral: REST
- mHealth (Active Comparator): Use of the "resilience" application on a smart phone to assess daily symptoms over 14 days and follow a self directed, symptom guided return to physical activity. Also Fitbit monitored.
  Interventions: Behavioral: mHEALTH
- Activity (Active Comparator): Low intensity activity regardless of symptoms using their Fitbit to measure said activity with goals (eg. 10,000 steps/ day.
  Interventions: Behavioral: ACTIVITY
- Both Activity and mHealth (Active Comparator): This group will receive both interventions and utilize the "SuperBetter" app. Interventions will be integrated by having research assistants support the subject to set and physical activity goals and milestones to the subject's pre-programmed general resilience goals in the SuperBetter© app (e.g. take a 30 min walk, march in place for 5 minutes, increase my step count by 2000 today, achieve 10,000 steps today).
  Interventions: Behavioral: ACTIVITY; Behavioral: mHEALTH

INTERVENTIONS:
Behavioral: REST — The REST group will be recommended to return to school and light physical and cognitive activity as soon as tolerated- but no sooner than 48 hrs post-injury per current consensus recommendations. Notifications from the Fitbit app will be turned off, and step goal will be set at 500, to minimize positive feedback and reminders from achievement of activity goals
  Arms: Rest
Behavioral: ACTIVITY — ACTIVITY group will be encouraged to engage in light to moderate physical activity with the goal of reaching 10,000 steps a day for one or more days during the first week. Subjects will be encouraged to engage in low-risk activities (e.g. walking). Subjects will be instructed to avoid activities that may increase risk of re-injury (e.g. bike riding, climbing, trampoline, sports). Fitbit notifications will be turned on and step goals will be set at 10,000. The simple goal of reaching 10,000 steps is clear to patients regardless of health literacy level, and real-time feedback provides continuous motivation.
  Arms: Activity; Both Activity and mHealth
Behavioral: mHEALTH — mHEALTH group will be instructed to download the SuperBetter© app. In addition to the pre-programmed general resilience goals, research assistants will help the subjects to set personal mental, social, and emotional rehabilitation goals and milestones for acute recovery from mTBI (e.g. return to school for ½ the day, have an improvement in symptoms). These goals/milestones will give the patient an opportunity to celebrate the achievement of improvement from mTBI with the goal of generating a positive contextual frame for recovery.
  Arms: Both Activity and mHealth; mHealth

SUMMARY:
The proposed interventions of this study will determine the ideal discharge recommendations related to activity

DETAILED DESCRIPTION:
The investigators will conduct a phase II factorial clinical trial . The clinical trial will determine the benefit of prescribed low-intensity physical activity, behavioral management, or both, versus standard rest in acute (24-48 hrs) (Moderate Traumatic Brain Injury (mTBI) patients presenting to the pediatric Emergency Department (ED). Low-intensity physical activity (i.e.10,000 steps/day) will be prescribed and monitored in the first week post-injury with an actigraph (Fitbit®). Behavioral management will be prescribed using a phone app referred to as mHealth (mobile Health, specifically SuperBetter©) that promotes mental, physical, social, and emotional resilience. This randomized clinical trial will have four treatment groups: 1) activity, 2) mHealth, 3) activity+mHealth, 4) rest. The primary study outcomes will be symptoms and recovery by 14 days. All subjects will be assessed via phone at 3-5 days and in person at 14 days. The secondary outcomes will be to determine the influence of interventions on comprehensive aspects of physiologic recovery and patient-centered outcomes; including symptoms at 3 days, neurocognitive, vestibular/ocular motor impairment at 14 days, pediatric quality of life measures, time to symptom resolution, and return to normal activity via phone survey at 1 and 2 months. The investigators will assess symptom, quality of life, and recovery outcomes based on treatment group assignment for all subjects and high-risk subjects.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mTBI in the past 72 hours

Exclusion Criteria:

* Patients having conditions otherwise which limit physical activity or neurocognitive assessment
* Do not have a smart phone
* History of brain surgery or past moderate/severe TBI within the last 6 months,
* Substance abuse,
* Major psychiatric condition under ongoing treatment with medications,
* Vestibular disorder,
* Cardiac condition,
* Unable to provide consent/assent
* Previous enrollment in the study

Ages: 11 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 237 (Actual)
Dates: Start 2019-06-11 (Actual); Primary Completion 2023-06-22 (Actual); Study Completion 2023-08-11 (Actual)

PRIMARY OUTCOMES:
Change in Post-Concussion Symptoms Scale (PCSS) | Day 0, Day 10-14
  Post-concussive symptoms at 14 days will be assessed using the Post-Concussion Symptom Scale (PCSS). We chose the 22-item PCSS as it is commonly used and would ensure consistency in longitudinal comparisons. The PI has validated PCSS administration via phone. The PCSS comprises 22 self-reported symptoms (e.g., dizziness headache) rated on a scale from 0 (none) to 6 (severe). PCSS score of ≤ 7 will be defined as symptom recovery. The PCSS takes 5 min to complete.
Change in Pediatric Quality of Life Measures (PedsQL) | Day 0, Day 10-14,
  We will assess health-related quality of life at 14 days using the PedsQL, a validated tool that has been used in healthy children and adolescents and those with acute and chronic health conditions. PedsQL has been demonstrated to show differences between subjects with persistent symptoms and those without up to 12 weeks post-concussion. The PedsQL measures have reliability and validity in assessing and comparing health-related quality of life scores between groups. They are agespecific and can be administered to parents and children and have been used to assess functional outcomes over time. The inventory includes 23 items rated from 0 (never) to 4 (almost always) and takes less than 5 min to complete.
Fitbit Flex 2 Actigraph | Day 0-14
  The Fitbit Flex 2 Actigraph will be distributed from the ED for all subjects in the study. Fitbit Actigraphs have been utilized in over 300 published studies. The Fitbit Flex 2 device to be worn by all subjects will provide objective activity metrics including measures of physical activity (e.g., number of steps per day, active minutes, distance traveled) and sleep (e.g., time to fall asleep, time sleeping, restless time). The Fitbit Flex 2 has a up to 5 days of battery life (device reminds subjects when battery life is low). The device 5 LEDs can be utilized to remind subjects to move, remind of current step goals, and celebrate when the goal is met. These features will be activated for subjects in the ACTIVITY groups. These data will be extracted directly from each device through Fitbit's API (Application Programming Interface. Allows devices to communicate with other select devices) system. These data will be collected in the first 14 days postinjury.

SECONDARY OUTCOMES:
Symptom Tracking Assessment for Concussion (STAC) application | Day 0-14
  The mobile application used in this study features an adaptive assessment of post-concussive symptoms utilizing the Post Concussive Symptom Survey (PCSS), which presents a narrow symptom list that adapts to focus on symptoms reported by the subject on previous assessments. Additional data to be collected will include: a report of cognitive and social activity, a subjective estimate of most active time of day (for validation against Fitbit data), times of day not wearing Fitbit, and the degree to which symptoms were exacerbated by activities. We have shown that the app is used by most subjects and that self-reported physical activity levels in this app show reductions similar to what we have seen with the Fitbit.
Immediate Post-Concussion Assessment and Cognitive Test (ImPACT) | Day 0, Day 10-14,
  The Immediate Post-Concussion Assessment and Cognitive Test (ImPACT) computerized test will be used to assess neurocognitive function. The ImPACT test assesses attention processes, visual working memory, verbal recognition memory, reaction time, visual processing speed, numerical sequencing ability, and learning. These modules are aggregated into four composite scores: verbal and visual memory, motor processing speed, and reaction time. The sensitivity of ImPACT is 81.9%, and the specificity is 89.4%. Research on the validation and test re-test reliability of ImPACT is reported elsewhere. The PI has validated ImPACT in the pediatric emergency department in several previous studies. The ImPACT test takes 30 min to complete (including the PCSS)
Vestibular/Ocular Motor Screen (VOMS) | Day 0, Day 10-14,
  We will assess vestibular/ocular motor impairment using the Vestibular/Ocular Motor Screen (VOMS) The VOMS assesses: 1) smooth pursuits, 2) horizontal and vertical saccades, 3) convergence, 4) horizontal and vertical vestibular ocular reflex and 5) visual motion sensitivity. Subjects verbally rate on a scale of 0 (none) to 10 (severe) changes in headache, dizziness, nausea and fogginess symptoms compared to their pre-assessment state following each VOMS assessment to assess symptom provocation. Convergence is assessed via symptom report and near point of convergence (NPC). NPC values > 5 cm are considered abnormal. The VOMS takes 5 min to administer.
Modified Balance Error Scoring System (mBESS) | Day 0, Day 10-14,
  We will assess balance using the modified Balance Error Scoring System (mBESS), a costeffective way to objectively assess balance. The test consists of three stance conditions (double leg, single leg, tandem) performed on firm flooring. In all stances, errors are recorded as the quantitative measurement of postural stability. Performance is scored by adding the error points according to the mBESS for each of the three trials. Trials are incomplete if subjects do not sustain the stance position for longer than 5 seconds. In this case, a standard maximum score of 10 is assigned for the trial. The mBESS takes 5 min to administer.
International Activity Questionnaire (IPAQ) | Day 0, Day 10-14, Day 30, Day 60
  Pre-injury activity level will be assessed in order to determine if discharge instructions lead to a decrease in post-injury activity level. To do this, we will utilize the International Activity Questionnaire (IPAQ). This is a validated tool to assess recall of average activity level and intensity over the preceding 7 days. It was chosen because it is brief and can be either self-administered or administered via structured phone interview. Activity levels can be expressed as categorical variables (Low, medium, high activity levels) or a continuous variable (MET-min/ week). We will also include the cognitive activity assessment used by Brown and colleagues. This measure assesses (on a scale of 1-4) the average level of cognitive activity including tests, reading, homework, texting, and video games during the past 7 days. The combined IPAQ and cognitive activity assessment take 5 min to complete.
Brief Symptom Inventory-18 (BSI-18) | Day 3-5, Day 30, Day 60
  The Brief Symptom Inventory (BSI) gathers patient reported data to assess psychological distress and psychiatric disorders. It tests three primary symptom dimensions (Depression, Anxiety, and Somatization) and is designed to assess changes throughout treatment. The BSI-18 asks 18 items are rated on a 5-point rating scale, 0 (Not at all) to 5 (Extremely). It is scored on the three primary symptoms dimensions and an overall Global Severity Index. Our research team has utilized the BSI-18 in the ED setting. The BSI-18 takes 4 minutes to complete.
Screen Time Assessment | Day 0 - 14
  Screen Media Use and Internet Use (Screens) REF
  Measures of screen time and internet use. Assess screen media use items:
  * Amount of time in screen use
  * Assess internet use
  * 5 items
  * 8 point scale (1 = definitely disagree to 8 = definitely agree) Primary metric = Mean scores hours of screen media use and internet use

CONTACTS AND LOCATIONS:
Overall Officials: Danny Thomas, MD, Principal Investigator — Medical College of Wisconsin
Locations (2):
- United States (2):
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
CoInvestigator on the study and the identified study teams for both Children's Hospitals in Milwaukee, WI (WI) and Pittsburgh, PA (Pennsylvania) will be involved in collecting and analyzing study data
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Throughout the described life of the study indicated earlier.
Access Criteria: Upon request.

REFERENCES:
- [Derived] Thomas DG, Erpenbach H, Smith CN, Hickey RW, Waltzman D, Haarbauer-Krupa J, Nelson LD, Patterson CG, McCrea M, Collins MW, Kontos AP. Impact of Early Activity and Behavioral Management on Acute Concussion Recovery: A Randomized Controlled Trial. J Pediatr. 2025 Aug;283:114596. doi: 10.1016/j.jpeds.2025.114596. Epub 2025 Apr 18. PMID 40254050
- [Derived] Eagle SR, Zynda AJ, Sandulli L, Hickey RW, Kegel NE, Nelson L, McCrea M, Collins MW, Okonkwo DO, Thomas DG, Kontos AP. The Role of Body Mass Index on Physical Activity, Symptoms, and Related Outcomes Following Pediatric Concussion. J Pediatr. 2025 Feb;277:114386. doi: 10.1016/j.jpeds.2024.114386. Epub 2024 Nov 1. PMID 39489284